CLINICAL TRIAL: NCT00110942
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Systemic AMG 108 in Subjects With Osteoarthritis (OA)
Brief Title: Treatment for Patients With Osteoarthritis (OA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20040166
Record Dates: First submitted 2005-05-16; First posted 2005-05-17 (Estimated); Last update posted 2008-06-23 (Estimated); Status verified 2008-06

CONDITIONS: Osteoarthritis
Keywords: Intra-articular; Osteoarthritis; OA; anakinra; Amgen
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Minor sub-study AMG 108 (Active Comparator): N = 15
  Interventions: Drug: Systemic AMG 108
- Minor sub-study placebo (Placebo Comparator): N = 15
  Interventions: Other: Placebo
- Main sub-study AMG 108 (Active Comparator): N = 73
  Interventions: Drug: Systemic AMG 108
- Main sub-study placebo (Placebo Comparator): N = 73
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Systemic AMG 108 — 300 mg SC AMG 108 Q4W for 3 doses
  Arms: Main sub-study AMG 108; Minor sub-study AMG 108
Other: Placebo — SC placebo injection Q4W for 3 doses
  Arms: Main sub-study placebo; Minor sub-study placebo

SUMMARY:
The purpose of this study is to evaluate the clinical benefit (change in Western Ontario and McMaster University Osteoarthritis Index [WOMAC] pain score) of AMG 108 (300 mg subcutaneously [SC] every 4 weeks) in subjects with OA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee OA as determined by American College of Rheumatology (ACR) criteria
* Pain defined by a level of greater than or equal to 30 mm on a 100 mm Visual Analogue Scale (VAS)
* If currently taking any over the counter nutritional supplements, must be on stable doses for greater than 2 months prior to screening
* If utilizing physical therapy, biomechanical devices or orthotic support, must have been using treatment or device for greater than or equal to 2 months prior to screening
* If currently or previously taking any non-prescribed supplement (e.g., glucosamine or chondroitin sulphate, shark cartilage, diacerein, soya extract, etc.) must be on stable doses for at least 2 months prior to screening
* If currently taking nonsteroidal anti-inflammatory drugs (NSAIDs), must be on stable doses for at least 2 months prior to screening
* Able to discontinue NSAIDs at least 5 half-lives (approximately 3 days) prior to Day 1
* Radiographic evidence of tibio-femoral compartment knee OA within 12 months of screening
* Signed written informed consent

Exclusion Criteria:

* Malignancy within the previous 5 years, except for basal cell or in situ cancer
* Significant hematologic disease - Active infection or history of recurrent or chronic infections
* Known diagnosis of HIV, hepatitis B, or hepatitis C infection
* Uncontrolled diabetes or cardiovascular disease and hypertension
* Inflammatory arthropathy including secondary OA
* Isolated OA of the patellofemoral joint (bi or tri-compartmental involvement are not exclusions)
* End-stage ("bone-on-bone") OA (Kellgren Lawrence score of 4)
* OA of the hip ipsilateral to the index knee - Total white cell count less than 2.0 x 10^9/L and/or platelet count less than 100 x 10^9/L observed within 1 month preceding screening
* Prior intra-articular (IA) injection of anakinra or experimental interleukin-1 (IL-1) inhibitor therapy - Concurrent treatment with SC anakinra
* Concurrent or recent (less than or equal to 1 month) use of experimental therapy
* Prior IA corticosteroid injection within 1 month of study
* Prior viscosupplement therapy within 3 months of study
* Contraindication(s) to IA injections
* Subjects who are pregnant or breast-feeding, or plan to become pregnant during the study
* Subject is not using adequate contraception
* Known allergy to E coli-derived products
* Unable to understand informed consent
* Concerns regarding subject's compliance with the protocol procedures
* Subject will not be available for follow-up assessment
* Active substance abuse

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2005-02; Primary Completion 2005-06 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC pain score | Week 6

SECONDARY OUTCOMES:
Change in WOMAC pain score | Week 12
Change in WOMAC composite score and function and stiffness index scores | Weeks 6 and 12
Achieving 50% or more improvement from Day 1 in the WOMAC | Weeks 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Cohen SB, Proudman S, Kivitz AJ, Burch FX, Donohue JP, Burstein D, Sun YN, Banfield C, Vincent MS, Ni L, Zack DJ. A randomized, double-blind study of AMG 108 (a fully human monoclonal antibody to IL-1R1) in patients with osteoarthritis of the knee. Arthritis Res Ther. 2011 Jul 29;13(4):R125. doi: 10.1186/ar3430. PMID 21801403
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/2004166.pdf